CLINICAL TRIAL: NCT03666390
Title: A Double-blind, Randomized-controlled Trial Using a Low Dose of Ketamine vs. Active Placebo in Treating Severe Depression and Suicide
Brief Title: Using a Low Dose of Ketamine vs. Active Placebo in Treating Severe Depression and Suicide
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 107-2314-B-075-063-MY3
Record Dates: First submitted 2018-09-09; First posted 2018-09-11 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Major Depressive Disorder
Keywords: treatment refractory depression; suicide; ketamine
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Suicide | interventions — Ketamine; Midazolam

STUDY DESIGN:
Intervention Model Description: 0.5mg/kg vs. active placebo (0.045mg/kg Midazolam)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.5mg/kg Ketamine (Experimental): Anesthesia
  Interventions: Drug: Ketamine
- 0.045mg/kg Midazolam (Active Comparator): Benzodiazepine
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — We will elucidate the exact efficacy of a low dose of ketamine infusion for the rapid anti-depression and anti-suicidal ideations.
  Other Names: Ketalar
  Arms: 0.5mg/kg Ketamine
Drug: Midazolam — We will elucidate the exact efficacy of a low dose of ketamine infusion for the rapid anti-depression and anti-suicidal ideations.
  Other Names: Dormicum
  Arms: 0.045mg/kg Midazolam

SUMMARY:
Depression and suicide are two leading mental health and public health issues in Taiwan. However, until now, the optimal treatment for refractory depression and suicide is still lacking. Previous USA studies suggested a low dose NMDA antagonist Ketamine infusion can significantly reduce depression and suicide. In our study, we firstly investigate the anti-suicide and anti-depressive effects of ketamine in Taiwan. If we can find the similar antidepressant and anti-suicide of ketamine in Taiwanese, this result will have a great influence in the current suicide and depression prevention programs.

DETAILED DESCRIPTION:
Depression and suicide are major issues of public health worldwide. However, there is time-lag for current available antidepressants to have therapeutic effective. In fact, if partial responses were also included, up to 50% of depressed patients showed little or no response to traditional antidepressant medication treatments. In addition, suicide is also a prevalent mental health problem worldwide and still has no optimal and effective treatment now. In Taiwan, the annual suicide rate increased gradually despite of the suicide prevention program. Ketamine, a kind of N-methyl-D-aspartate receptor (NMDAR) antagonist, is a FDA-approved anesthetic agent. One single sub-anesthesia dose of ketamine infusion can rapidly improve refractory depression without side effects of dependence, and its antidepressant effects have been proved by some double-blind and randomized controlled trials in other countries. However, it has not been investigated and validated in Han Chinese population. The mechanism of rapid antidepressant effects is still unknown. Besides, much less studies assessed the anti-suicide efficacy of a low dose of ketamine infusion.

Under the support of NSC 101-2314-B-010-060 and NSC 101-2314-B-010-061, we finished the study of a single dose ketamine infusion in the treatment of refractory major depression (TRD) using a double blind randomized placebo-controlled fashion. Three groups with each 24 patients of TRD received 0.5mg/kg, 0.2mg/kg and placebo (PBO) respectively. The primary outcome assessed by MADRS and HAMD depression ratings disclosed about 40~45% response. Also, a single low dose of ketamine could reduce approximately 50% suicide-related symptoms based on the subanalysis of ketamine treatment efficacy for specific suicide item.

In current study, we plan to recruit 48 subjects of TRD within two years in double-blind, randomized - controlled fashion with each year 24 subjects, who will receive 0.5mg/kg vs. active placebo (0.045mg/kg Midazolam) equally. Mood symptom changes by MARDRS and HAMD ratings, suicide scales, and impulsivity and loneliness scales will be conducted at different time points from baseline to the 14th day. We will elucidate the exact efficacy of a low dose of ketamine infusion for the rapid anti-depression and anti-suicidal ideations. If it is successful, it would be able to generalize to benefit for the huge population of Chinese in the world.

ELIGIBILITY:
Inclusion Criteria:

1. Major depression including unipolar and bipolar depression, according to DSM-IV criteria and MINI (MiniInternational Neuropsychiatric Interview;MINI) diagnostic interview.
2. Age ≧ 20y/o < 65 y/o
3. voluntary patients with signed informed consent proved by institutional review board (IRB)

Exclusion Criteria:

1. Major medical conditions (e.g., head injury, epilepsy, severe renal diseases and cancer).
2. Other axis I psychiatric disorders such as schizophrenia, delusional disorder, organic brain syndrome, and dementia.
3. Pregnancy.
4. Substance abuse in previous 6 months such as cocaine, marijuana, opium, ketamine, PCP (phencyclidine)。
5. Current use of NMDA receptor antagonist (Amantadine, Rimantadine, Lamotrigine, Memantine, Dextromethorphan)
6. Alcohol abuse / dependence within 6 months.
7. Attempt suicide in hospital.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-09-10 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction rate of suicide symptom | 4 hours, 1 day, 2 days, 3 days, 4 days, 5 days, 6 days, 7 days, 14 days.
  Reduction rate of suicide symptom postinfusion of ketamine

SECONDARY OUTCOMES:
Reduction rate of depression symptom | 4 hours, 1 day, 2 days, 3 days, 4 days, 5 days, 6 days, 7 days, 14 days.
  Reduction rate of depression symptom post-infusion of ketamine

CONTACTS AND LOCATIONS:
Overall Officials: Mu-Hong Chen, M.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided